CLINICAL TRIAL: NCT02743039
Title: The Northwestern University Two-Generation Study of Parent and Child Human Capital Advancement
Acronym: NU2Gen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Teresa Eckrich Sommer, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00201886
Record Dates: First submitted 2016-04-07; First posted 2016-04-19 (Estimated); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Children; Parents
Keywords: Low income; Education; Poverty; Children; Parents; Head Start

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CareerAdvance® (Experimental): CareerAdvance® provides education, career coaching, and soft-skills training for parents while their children attend Head Start programs.
  Interventions: Behavioral: CareerAdvance®
- Control Standard of CAP (No Intervention): No assignment to participate in the CareerAdvance® program, but given community referrals and resources

INTERVENTIONS:
Behavioral: CareerAdvance® — CareerAdvance® is a dual-generation program providing education, career coaching, and soft-skills training for parents while their children attend CAP Tulsa's Head Start programs.
  Arms: CareerAdvance®

SUMMARY:
The Northwestern University Two-Generation Child and Family Outcomes Study (NU2Gen) of the Community Action Project of Tulsa County's (CAP Tulsa's) CareerAdvance® program examines the effects of CareerAdvance® on parent and child human capital outcomes (e.g., child academic achievement, parent educational advancement and certification, and psychological and family functioning), and (2) explore mechanisms that might give rise to program effects (e.g., home language environment; coping, balance, and stress; and parent and academic and career identity).

DETAILED DESCRIPTION:
The Northwestern University Two-Generation Study (NU2Gen) of Parent and Child Human Capital Advancement is funded through Community Action Project of Tulsa County's (CAP Tulsa) Health Profession Opportunity Grant (HPOG II) from the Administration for Children and Families and through the HPOG II University Partnership grant. The federal awards support the implementation of CareerAdvance®, a workforce training and career employment program for parents living in Tulsa, Oklahoma and the surrounding communities, as well as our Northwestern-based research project.

CareerAdvance® provides education and training, career coaching, and other supportive services for parents while their children attend CAP Tulsa-run Head Start programs, other Tulsa-area public preschool programs, and Tulsa-area K-12 public schools. The explicit goal of the program is to promote the economic self-sufficiency and well-being of low-income families across generations.

The evaluation is composed of two parts: the Two-Generation Human Capital Outcomes Study and the Two-Generation Explanatory Mechanisms Study. Through parent surveys and parent and child administrative data we will examine the effects of CareerAdvance® on parent and child human capital outcomes (e.g., child academic achievement, parent educational advancement and certification, and psychological and family functioning). Using innovative measurement tools (e.g. Language Environment Analysis (LENA)) along with parent and child focus groups and interviews, we will also explore mechanisms that might give rise to program effects (e.g., home language environment; coping, balance, and stress; and academic and career identities). Participants will actively take part in the study for three years and we will collect child administrative data for study parents' children until they turn 18 years old or graduate high school, whichever occurs last. Current funding for NU2Gen is through September 2020.

ELIGIBILITY:
Inclusion Criteria:

* Applicants to CAP Tulsa's CareerAdvance® program under the HPOG II evaluation study, including participants who are randomly assigned not to participate in CareerAdvance® by the HPOG II evaluation study.

Exclusion Criteria:

* Not proficient in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2016-04; Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Parent's employment | Year 2
  We expect higher rates of employment
Parent's healthcare sector employment | Years 1 and 2
  We expect higher rates of employment in the healthcare sector
Parent's income | Year 2
  We expect higher income
Parent's income | Year 1
  We expect lower income
Parent's healthcare training certification | Years 1 and 2
  We expect higher rates of healthcare training certification and credentialing
Child's academic achievement | Year 2
  We expect higher levels of academic achievement
Child's attendance | Years 1 and 2
  We expect higher rates of school attendance
Child's grade promotion | Years 1 and 2
  We expect higher rates of grade promotion

SECONDARY OUTCOMES:
Parent's depression | Year 2
  We expect less depression; Beck Depression Inventory-II (BDI-II; Beck, Steer, & Brown, 1996)
Parent's optimism | Year 2
  We expect increased optimism; Revised Life Orientation Test (LOT-R; Scheier, Carver, & Bridges, 1994)
Parent's work-family balance | Year 2
  We expect better work-family balance; Fragile Families Study; CAP Family Advancement Study (NU)
Parenting stress | Year 1
  We expect stable or increased parenting stress; Aggravation in Parenting Questionnaire (APQ; Cooper et al., 2009); Fragile Families Study
Parent's perceived stress | Year 1
  We expect stable or increased perceived stress; Perceived Stress Scale (PSS; Cohen & Williamson, 1988)
Parent's hope/goal efficacy | Year 2
  We expect higher levels of hope/goal efficacy; State Hope Scale (Snyder et al., 1996)
Parent's social capital | Year 2
  We expect higher social capital; Willingness to ask for/offer help (Adapted from the Boston Non-Profit Organizations Study survey; Tran, Graif, Jones, Small, & Winship, 2013)
Child adaptive skills | Year 2
  We expect an increase in child adaptive skills; Social Skills Improvement System (SSIS-RS; Gresham & Elliott, 2008)
Home language environment | Year 2
  We expect an increase in positive home language environment factors (e.g., books, reading time, learning activities) and a decrease in negative home language environment factors (e.g., television, video games/computer time, phone); Language Environment Analysis (LENA) system
Time use | Year 2
  We expect improved time use in the home; LENA Time Diary (Northwestern University, 2017)
Routines | Year 2
  We expect more stable routines in the home
Child emotional and behavior problems | Year 1
  We expect stable or increased child behavior problems; Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2000)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa E Sommer, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University, Evanston, Illinois
  - Community Action Project of Tulsa County, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Study description via website — https://sites.northwestern.edu/nu2gen/sample-page/current-studies/community-based/